CLINICAL TRIAL: NCT03917667
Title: Sarcopenia in Acute Care Patients: Protocol for Sarcopenia 9+
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of Geriatry Department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Sarcopenia 9+
Record Dates: First submitted 2019-04-03; First posted 2019-04-17 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Sarcopenia
Keywords: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric patients: Patients aged 70 years and older who are admitted to the acute care geriatric units.
  Interventions: Diagnostic Test: EWGSOP2

INTERVENTIONS:
Diagnostic Test: EWGSOP2 — EWGSOP2 criteria (Writing Group for the European Working Group on Sarcopenia in Older People 2) will be followed to determine the diagnosis of sarcopenia, considered as a dichotomous variable -yes/no- in presence of low grip strength + low muscle mass + low gait speed.

SUMMARY:
Sarcopenia is a disease characterized by progressive and generalized loss of skeletal muscle mass and strength, and is related to worse clinical outcomes, physical impairment, and mortality in all healthcare settings. This nutrition-related syndrome is a reversible condition, and can be effectively counteracted by exercise and nutritional support.

The prevalence of sarcopenia varies widely depending on the criteria, methods, and cut-off points used for its assessment. Although the European Working Group on Sarcopenia in Older People (EWGSOP) recommended assessing sarcopenia in geriatric patients in all care settings, few studies addressing hospitalized older patients have been carried out, mainly due to the characteristics of acute healthcare settings and their in-patients and because the criteria used are difficult to carry out there. Therefore, this condition remains under-recognized in the setting where this disease is likely to be more present.

Sarcopenia is expected to be a major healthcare problem in the upcoming years in Europe so, in response to this claim for Public Health Action, the European Union Geriatric Medicine Society founded the Special Interest Group (SIG) on sarcopenia that has taken the lead of bridging the gaps between clinical and research in sarcopenia field, in line with the Conference on Frailty and Sarcopenia Research Task Force, and the World Health Organization's strategies to promote Optimal Aging. This goal of SIG on sarcopenia by EuGMS is being carried out by promotion of collaboration among International scientific societies and institutions; they have recently launched the Revised European consensus on definition and diagnosis (EWGSOP2), the SARCUS project on ultrasound for sarcopenia assessment in European countries, and the first International Registry of patients with sarcopenia.

This study aims to provide an overview of sarcopenia assessment older patients hospitalized in acute-care geriatric units.

This is a longitudinal, prospective, observational study in consecutive hospitalized patients in the CHU Brugmann Hospital.

This study has 5 objectives :

1. To determine prevalence of sarcopenia among hospitalized patients in CHU Brugmann.
2. To determine incidence of sarcopenia during the hospital stay.
3. To identify risk factors for the development of sarcopenia at the time of admission and during hospitalization.
4. To assess sarcopenia as a risk factor for clinical adverse outcomes during hospitalization (hospital-acquired infections, falls, delirium, longer length-of-stay, disability, and mortality).
5. To assess sarcopenia as a risk factor for clinical adverse outcomes post-discharge (institutionalization, hospitalizations, falls, disability, and mortality) at 3- and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 70 years and older who are admitted to the acute care geriatric units of the CHU Brugmann Hospital.

Exclusion Criteria:

* Hip or lower limbs fractures, amputations,
* Terminally ill patients admitted for palliative care,
* Neurological patients with hemiplegia or stroke limiting the walking evaluation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 70 years and older who are admitted to the acute care geriatric units of the CHU Brugmann Hospital. This may include acute medical conditions or chronic disease decompensation; patients are eligible for referral to acute geriatric units due to medical diseases, such as urinary tract infections, respiratory tract infections, pneumonia, coronary heart diseases, atrial fibrillation, congestive heart failure, stroke, delirium, electrolyte disturbances, kidney disease, cancer, etc...
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia at hospital admission | 72 hours
  Prevalence of sarcopenia at hospital admission. A prevalent case of sarcopenia will be considered if a patient fulfills the EWGSOP2 at admission
Incidence of sarcopenia between admission and discharge | Up to 20 days
  A incident case of sarcopenia will be considered if a patient that do not fulfill EWGSOP2 diagnostic criteria at admission, fulfills the diagnostic criteria at discharge (diagnosis will be considered as a dichotomous variable -yes/no-).
Occurence of risk factors | Up to 20 days
  Presence of at least one risk factor involved in the development of sarcopenia during hospitalization. Risk factors defined as: bed immobilization, denutrition, loss of autonomy, cognitive troubles, depression, mobility loss.
Occurence of adverse events | Up to 20 days
  Presence of at least one adverse event of the following list: Falls, Fracture, Delirium, Aspiration, Pneumonia, Urinary tract infection, Gastrointestinal infection, Sepsis, Gastrointestinal bleeding, Decubitus ulcer (Bed sores), Deep vein thrombosis, Pulmonary embolism, Arrythmia, Stroke, Myocardial infarction, Cardiopulmonary arrest, Death, Date of death, Hospital re-admission, Institutionalisation, Emergency Department visits.
Occurence of adverse events | 3 months after hospital discharge
  Presence of at least one adverse event of the following list: Falls, Fracture, Delirium, Aspiration, Pneumonia, Urinary tract infection, Gastrointestinal infection, Sepsis, Gastrointestinal bleeding, Decubitus ulcer (Bed sores), Deep vein thrombosis, Pulmonary embolism, Arrythmia, Stroke, Myocardial infarction, Cardiopulmonary arrest, Death, Date of death, Hospital re-admission, Institutionalisation, Emergency Department visits.
Occurence of adverse events | 1 year after hospital discharge
  Presence of at least one adverse event of the following list: Falls, Fracture, Delirium, Aspiration, Pneumonia, Urinary tract infection, Gastrointestinal infection, Sepsis, Gastrointestinal bleeding, Decubitus ulcer (Bed sores), Deep vein thrombosis, Pulmonary embolism, Arrythmia, Stroke, Myocardial infarction, Cardiopulmonary arrest, Death, Date of death, Hospital re-admission, Institutionalisation, Emergency Department visits.

CONTACTS AND LOCATIONS:
Overall Officials: Murielle Surquin, MD, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - UZ Gent, Ghent

IPD SHARING:
Plan to Share IPD: No